CLINICAL TRIAL: NCT00062530
Title: Development of an Oral Prime-Boost AIDS Vaccine to Elicit Broadly Neutralizing Antibodies Against HIV-1
Brief Title: Safety of an Oral HIV Vaccine in HIV Uninfected Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Greg K. Lewis, PhD, University of Maryland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P01AI047490 (NIH); P01AI047490 (NIH)
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: AIDS; HIV seronegativity; HIV preventive vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

ARMS (1):
- 1 (Experimental): All participants will receive oral vaccine at study entry, although dosage will vary
  Interventions: Biological: SCBaL/M9

INTERVENTIONS:
Biological: SCBaL/M9 — Oral recombinant Salmonella typhi HIV-1 gp120 vaccine

SUMMARY:
This study will test the safety of and immune response to an oral HIV vaccine in healthy volunteers. The vaccine in this study uses a weakened bacterium called Salmonella typhi to deliver an HIV gene into the body through the mouth. The body then produces an HIV protein from the gene; this protein stimulates an anti-HIV immune response. The vaccine contains only one of the many substances that HIV needs to make more copies of itself, so the vaccine itself cannot cause HIV or AIDS.

DETAILED DESCRIPTION:
The transmission of HIV-1 by both sexual and parenteral routes makes it likely that a successful preventive vaccine against this virus will need to induce protective immunity in both mucosal and systemic compartments. The long-term objective of this program is to develop an HIV-1 vaccine that elicits protective immunity in both the mucosal and systemic compartments.

The study will evaluate the safety and immunogenicity of an oral recombinant Salmonella typhi HIV-1 gp120 vaccine (SCBaL/M9) in healthy human volunteers. This will be the first study in volunteers to use an intracellular bacterium to deliver a recombinant vector vaccine mucosally. The study will also develop an Env immunogen that elicits a broader spectrum of neutralizing antibodies than gp120 and that can be delivered by Salmonella typhi or as a soluble protein immunogen.

This is a Phase I dose-escalation study of two vaccine components that will be combined in a larger prime-boost protocol should the desired safety endpoints be obtained. Both components use a conformationally constrained gp120 that expresses epitopes recognized by broadly neutralizing antibodies. The priming immunogen will be the conformationally constrained gp120 gene delivered orally by live attenuated Salmonella typhi. The boosting immunogen will be a soluble subunit protein comprised solely of the conformationally constrained gp120.

All participants in this study will receive the vaccine. Participants will be randomized to different vaccine doses. Participants will have eight study visits over 20 weeks. Study visits will include brief medical interview, physical exam, blood and urine tests, and counseling on avoiding HIV infection and pregnancy. Participants will be tested for HIV infection 3 times during the study.

ELIGIBILITY:
Inclusion Criteria

* HIV uninfected
* Low risk sexual behavior
* Negative for Hepatitis B surface antigen
* Negative for Hepatitis C viral sequences and antibody
* Availability for follow-up for planned duration of the study (12 months)
* Acceptable methods of contraception

Exclusion Criteria

* Receipt of HIV vaccines or placebo in a previous HIV vaccine trial
* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications
* History of cancer unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure
* Medical or psychiatric condition or occupational responsibilities which preclude compliance with the protocol
* History of suicide attempts, recent suicidal ideation, or psychosis
* High risk behavior for HIV infection as determined by screening questionnaire
* History of injection drug use within 12 months of study entry
* Live attenuated vaccines within 60 days of study entry. Medically indicated killed or subunit vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 2 weeks away from HIV immunizations.
* Use of experimental agents within 30 days of study entry
* Receipt of blood products or immunoglobulin within 6 months of study entry
* Active syphilis
* Active tuberculosis
* History of anaphylaxis or serious adverse reactions to vaccines
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension)
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)

PRIMARY OUTCOMES:
Safety, as judged by the lack of an immune response to CD4 epitopes or other significant adverse events as defined by the HVTN toxicity tables | Throughout study

SECONDARY OUTCOMES:
Neutralizing antibody response against HIV-1 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: George K. Lewis, PhD, Principal Investigator — Univesity of Maryland
Locations (1):
- Institute of Human Virology, Baltimore, Maryland, United States